CLINICAL TRIAL: NCT06797427
Title: An Open-label, Prospective, Randomised, Cross-over Trial to Assess the Pharmacokinetics of an Amorphous Formulation of Sorafenib in Mesoporous Magnesium Carbonate (DPH001) Compared to Nexavar® (sorafenib) in Healthy Volunteers
Brief Title: A Study to Assess the Pharmacokinetics of Sorafenib in Mesoporous Magnesium Carbonate (DPH001) Compared to Nexavar® (sorafenib) in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Disruptive Pharma (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPH001-01; 2024-514496-18 (EudraCT Number)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: PK study; Sorafenib; Hepatocellular carcinoma; MMC; Amorphous formulation; Mesoporous magnesium carbonate; Absorption; Bioavailability; Drug delivery; Kinase inhibitors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single dose of Nexavar sorafenib (Active Comparator): 1 dose of 200 mg sorafenib as Nexavar®, film-coated tablets for oral administration, in a fasted state. IMP administrations (dosing) will be separated by wash-out periods of at least 14 days
  Interventions: Drug: Nexavar (Sorafenib)
- Singel dose of DPH001 (Experimental): 1 dose of 100 mg sorafenib as DPH001, HPMC capsuls for oral administration, in a fasted state. IMP administrations (dosing) will be separated by wash-out periods of at least 14 days
  Interventions: Drug: DPH001

INTERVENTIONS:
Drug: DPH001 — 100 mg
  Arms: Singel dose of DPH001
Drug: Nexavar (Sorafenib) — 200 mg
  Arms: Single dose of Nexavar sorafenib

SUMMARY:
The study aims to assess the pharmacokinetics and safety of DPH001, an amorphous formulation of sorafenib, compared to Nexavar® in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, prospective, randomized, cross-over, single-center trial designed to evaluate the bioavailability, safety, and tolerability of DPH001 compared to Nexavar® in healthy male participants and healthy female participants of non-childbearing potential. The objective of the study is to compare the pharmacokinetics (PK) of sorafenib after the administration of 100 mg DPH001 vs. after the administration of 200 mg Nexavar®. After being informed of the study and potential risks, all subjects given written informed consent will undergo a screening to determine eligibility for study entry. Participants will receive, in a randomized order, 1 dose of 100 mg DPH001, and 1 dose of 200 mg Nexavar®, all in a fasted state. IMP administrations will be separated by wash-out periods of at least 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial, including consenting to the planned restrictions during the trial.
2. Healthy male or female participant aged 18 to 65 years, inclusive.
3. Body mass index (BMI) ≥18.5 and ≤30.0 kg/m2 at the time of the screening visit.
4. Medically healthy participant without abnormal clinically significant medical/surgical history, physical findings, vital signs, ECG, and laboratory values at the time of the screening visit, as judged by the Investigator.
5. Female trial participants: Only female participants of non-childbearing potential will be considered eligible for participation. Female participants of non-childbearing potential are defined as:

   * pre menopausal females who have undergone hysterectomy and/or bilateral salpingectomy and/or bilateral oophorectomy,
   * post menopausal females, defined as having undergone at least 12 months of amenorrhea. In questionable cases a blood sample with detection of follicle stimulating hormone (FSH) >25 IU/L will be confirmatory.

Male trial participants: Male participants must be willing to use condoms during sexual intercourse to prevent pregnancy and/or the drug exposure of a partner from the first IMP administration at Visit 2 and until 3 months after the last IMP administration at Visit 12.

In addition, any female partner of a male participant who is of childbearing potential must use contraceptive methods with a failure rate of <1%/year to prevent pregnancy from at least 2 weeks prior to the first administration of IMP to 3 months after the last administration of IMP.

The following are considered highly effective methods of contraception:

* combined (oestrogen and progestogen-containing) or progestogen-only hormonal contraception associated with the inhibition of ovulation (oral, transdermal, intravaginal, injectable, or implantable),
* intrauterine device (IUD) or intrauterine hormone-releasing system (IUS).

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the (first) administration of IMP.
3. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the trial.
5. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or HIV antigen and antibodies.
6. After 10 minutes supine rest at the screening visit, any vital signs values outside the following ranges:

   * systolic blood pressure: <90 or ≥140 mmHg, or
   * diastolic blood pressure <50 or ≥90 mmHg, or
   * pulse <40 or ≥90 bpm.
7. A mean QTcF interval of ≥450 ms at screening or a family history of long QT syndrome, as judged by the Investigator.
8. Abnormal ECG morphology at screening, including abnormality in PR and/or QRS intervals, as well as signs of bundle branch block (BBB), as judged by the Investigator.
9. History of cardiac arrhythmias or palpitations, including ectopic heart beats and/or extra systoles (premature ventricular contractions), as judged by the Investigator.
10. Hepatic dysfunction, defined as serum transaminase (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) levels above the upper limit of normal (ULN) at screening, if considered clinically significant by the Investigator.
11. Any other clinically relevant abnormalities in clinical chemistry, haematology, and coagulation parameters from safety laboratory tests at screening, at the discretion of the Investigator.
12. History of severe reaction, including allergy/hypersensitivity, to drugs with a similar chemical structure, class, or mechanism of action to sorafenib, and/or reaction to any drug that led to significant morbidity, as judged by the Investigator.
13. History of or ongoing major depressive disorder (MDD) and/or any history of suicidal ideation (i.e., active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent), at the discretion of the Investigator.
14. Regular use of any prescribed or non-prescribed medications, at the discretion of the Investigator, including antacids, analgesics, antibiotics, anticoagulants, non-steroidal anti-inflammatory drugs, herbal remedies, vitamins, and mineral, within 2 weeks prior to the first planned IMP administration at Visit 2, except the following:

    * Prescribed and stable treatment with any hormone replacement therapy (HRT).
    * Occasional intake of paracetamol (maximum 2000 mg/day for a maximum of 3 consecutive days and not exceeding 3000 mg/week).
    * Nasal decongestants without cortisone, antihistamine, or anticholinergics for a maximum of 10 days.
15. Planned treatment or treatment with another investigational drug within 3 months prior to Visit 2. Participants consented and screened but not dosed in previous phase I trials will not be excluded.
16. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times/week before the screening visit will be allowed.
17. Positive test result for drugs of abuse or alcohol at screening.
18. History or manifestation at screening of drug abuse, alcohol abuse and/or excessive intake of alcohol, as judged by the Investigator.
19. History of, or current use, of anabolic steroids, as judged by the Investigator.
20. Excessive caffeine consumption defined by a daily intake of >5 cups (1 cup = approximately 240 mL) of caffeine-containing beverages, as judged by the Investigator.
21. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the last 3 months prior to screening.
22. The Investigator considers the participant unlikely to comply with trial procedures, restrictions, and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
To compare the AUC (0-6h) of sorafenib after the administration of 100 mg DPH001 vs. 200 mg Nexavar® in fasted conditions. | From administration of study drug until 4 days
  Blood samples will be collected in order to calculate a PK-profile. Area under the plasma concentration vs. time curve (AUC) from time 0 to 6 hours (AUC0 6h).
To compare the AUC (0-72 h) of sorafenib after the administration of 100 mg DPH001 vs. 200 mg Nexavar® in fasted conditions. | From administration of study drug until 4 days
  Blood samples will be collected in order to calculate a PK-profile. Area under the plasma concentration vs. time curve (AUC) from time 0 to 72 hours (AUC 0-72h).
To compare the AUC (inf) of sorafenib after the administration of 100 mg DPH001 vs. 200 mg Nexavar® in fasted conditions. | From administration of study drug until 4 days
  Blood samples will be collected in order to calculate a PK-profile. Area under the plasma concentration vs. time curve (AUC) from time 0 extrapolated to infinity (AUCinf).
To compare the Cmax of sorafenib after the administration of 100 mg DPH001 vs. 200 mg Nexavar® in fasted conditions. | From administration of study drug until 4 days
  Blood samples will be collected in order to calculate a PK-profile. Maximum observed plasma concentration (Cmax).
To compare the Tmax of sorafenib after the administration of 100 mg DPH001 vs. 200 mg Nexavar® in fasted conditions. | From administration of study drug until 4 days
  Blood samples will be collected in order to calculate a PK-profile. Time to Cmax (Tmax).

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events assessed by frequency. | From administration of study drug until end of trial (period 2 day 8).
  Number of events. Descriptive individual data.
Number of subjects with treatment-related adverse events assessed by seriouness. | From administration of study drug until end of trial (period 2 day 8).
  The seriousness of events. Descriptive individual data.
Number of subjects with treatment-related adverse events assessed by intensity. | From administration of study drug until end of trial (period 2 day 8).
  The intensity of events. Descriptive individual data.
Number of subjects with treatment-related adverse events assessed by relationship to study treatment. | From administration of study drug until end of trial (period 2 day 8).
  The relationship to study treatment. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the systolic blood pressure. | From administration of study drug until end of trial (period 2 day 8).
  Measured in mmHg, supine position after 10 minutes rest. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the diastolic blood pressure. | From administration of study drug until end of trial (period 2 day 8).
  Measured in mmHg, supine position after 10 minutes rest. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QRS. | From administration of study drug until end of trial (period 2 day 8).
  Measured in ms, supine position after 10 minutes rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QT. | From administration of study drug until end of trial (period 2 day 8).
  Measured in ms, supine position after 10 minutes rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter PQ/PR. | From administration of study drug until end of trial (period 2 day 8).
  Measured in ms, supine position after 10 minutes rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter QTcF. | From administration of study drug until end of trial (period 2 day 8).
  Measured in ms, supine position after 10 minutes rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the ECG parameter heart rate. | From administration of study drug until end of trial (period 2 day 8).
  Measured in ms, supine position after 10 minutes rest using an ECG machine. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the clinical chemistry parameters. | From administration of study drug until end of trial (period 2 day 8).
  Blood samples for analyzing hematology parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the hematology parameters. | From administration of study drug until end of trial (period 2 day 8).
  Blood samples for analyzing hematology parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the coagulation parameters. | From administration of study drug until end of trial (period 2 day 8).
  Blood samples for analyzing hematology parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the head. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the eyes. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the ears. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the nose. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the throat. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the skin. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the thyroid. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the neurological. | From administration of study drug end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the lungs. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the cardiovascular. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the abdomen (liver and spleen). | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the lymphnodes. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the physical examination of the extremities. | From administration of study drug until end of trial (period 2 day 8).
  Physical examination. Descriptive individual data.
Number of subjects with treatment-related adverse events assessed by frequency. | From administration of study drug until 72 hours.
  Number of events. Descriptive individual data.
Number of subjects with treatment-related adverse events assessed by seriouness. | From administration of study drug until 72 hours.
  The seriousness of events. Descriptive individual data.
Number of subjects with treatment-related adverse events assessed by intensity. | From administration of study drug until 72 hours.
  The intensity of events. Descriptive individual data.
Number of subjects with treatment-related adverse events assessed by relationship to study treatment. | From administration of study drug until 72 hours.
  The relationship to study treatment. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the clinical chemistry parameters. | From administration of study drug until 72 hours.
  Blood samples for analyzing hematology parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the hematology parameters. | From administration of study drug until 72 hours.
  Blood samples for analyzing hematology parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.
Number of subjects with a clinical significant change from baseline in the coagulation parameters. | From administration of study drug until 72 hours.
  Blood samples for analyzing hematology parameters will be collected through venepuncture or an indwelling venous catheter. Descriptive individual data.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Schultze, MD, Principal Investigator — Clinical Trial Consultants (CTC), Dag Hammarskjölds väg 10B, 752 37 Uppsala, Sweden
Locations (1):
- Clinical Trial Consultants (CTC), Dag Hammarskjölds väg 10B, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No